CLINICAL TRIAL: NCT06214091
Title: Safety and Efficacy of Early Gastrointestinal Decompression for Patients With Acute Severe Ischemic Stroke
Brief Title: Gastrointestinal Decompression in Stroke
Acronym: EAGER-ASSIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Jiayue Ding, Principle investigator, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EAGER-ASSIST-1
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Stomach Acidity; Pulmonary Infection; Gastrointestinal Decompression
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrointestinal decompression group (Experimental)
  Interventions: Procedure: Gastrointestinal decompression
- Control group (Placebo Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Gastrointestinal decompression — Gastric tube is inserted within 24-hour severe ischemic stroke attack; gastrointestinal decompression is performed for 48 hours.
  Arms: Gastrointestinal decompression group
Procedure: Control — Gastric tube is inserted within 24-hour severe ischemic stroke attack.
  Arms: Control group

SUMMARY:
Acute severe ischemic stroke is a life-threatening subtype of stroke. Due to stress ulcer and gastric reflux in acute stage, patients with severe ischemic stroke are always complicated with stomach bleeding and pulmonary infections, resulting in poor prognosis and even death. Reducing stomach acidity and avoiding gastric reflux play a pivotal role on controlling serious complications after austere ischemic attack. Gastrointestinal decompression is an cheap, safe, effective and acknowledgemented strategy for treating stomach bleeding and preventing gastric reflux in clinical settings. Early gastrointestinal decompression seems to be an available method to reduce stomach acidity and avoid gastric reflux after severe ischemic stroke. Therefore, we aimed to evaluate the safety and efficacy of early gastrointestinal decompression in patients with acute severe ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* severe AIS, including NIHSS score>20 in dominant hemisphere infarction, or NIHSS score>15 in non-dominant hemisphere infarction, or NIHSS consciousness score >1; · massive infarction, characterized by infarction area larger than 1/3 of the effected middle cerebral artery territory and/or the cerebellum territory presented in admitted computed tomography (CT) or MRI
* onset-to-needle time within 24 hours
* prestroke modified Ranking scales (mRS)≤1
* sign the informed consent.

Exclusion Criteria:

* Recent respiratory infection and/or gastrointestinal bleeding
* austere diseases such as tumors and dyscrasia
* intention to undergo emergency thrombectomy
* pregnant women or nursing mother
* contraindication for gastric tubes
* participating in other clinical trials within previous 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
90-day Death | 90 days
  Death rate at 90 days

SECONDARY OUTCOMES:
90-day mRS | 90 days
  mRS at 90 days
90-day Barthel scores | 90 days
  Barthel scores at 90 days
30-day mRS | 30 days
  mRS at 30 days
30-day Barthel scores | 30 days
  Barthel scores at 30 days

IPD SHARING:
Plan to Share IPD: Undecided